CLINICAL TRIAL: NCT05959811
Title: Meridian Yoga on Chemotherapy-induced Peripheral Neuropathy in Breast Cancer Patients
Acronym: CIPN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMUH112-REC3-077
Record Dates: First submitted 2023-06-20; First posted 2023-07-25 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: CIPN - Chemotherapy-Induced Peripheral Neuropathy; Breast Cancer
Keywords: yoga; CIPN; meridian energy
MeSH Terms: conditions — Breast Neoplasms | interventions — Yoga

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- meridian yoga (Experimental): 60 minutes yoga ,twice a week for 8 weeks
  Interventions: Other: yoga
- usual care group (No Intervention): 8 weeks of general care

INTERVENTIONS:
Other: yoga — 60 minutes yoga practice ,twice a week for 8 weeks
  Arms: meridian yoga

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN) is a common side effect in breast cancer patients with completion of chemotherapy, and that is characterized by associated clinical symptoms such as pain, tingling, numbness, and paresthesia etc. CIPN also interferes with patients' functions of daily living and leads to chronic functional decline and a reduced quality of life. Meridian yoga is beneficial to the treatment of patients with peripheral neuropathy and the improvement of their quality of life.

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy (CIPN) is a common side effect in breast cancer patients with completion of chemotherapy, and that is characterized by associated clinical symptoms such as pain, tingling, numbness, and paresthesia etc. CIPN also interferes with patients' functions of daily living and leads to chronic functional decline and a reduced quality of life. Meridian yoga is beneficial to the treatment of patients with peripheral neuropathy and the improvement of their quality of life.

Therefore, the aim of this study was to evaluate the efficacy of meridian yoga for CIPN in breast cancer patients. The investigators designed a clinical randomized controlled trial in which 80 patients with CIPN were equally divided into a control group (8 weeks of general care) and a treatment group (general care plus 16 times yoga interventions for 8 weeks). The assessment time was before (vision 1) and at the completion of 8 weeks of Meridian yoga treatment (vision 2). The primary outcome was the change in scores of the neuropathic pain scale (Chinese version). The secondary outcome was to the changes of meridian energy [Meridian Energy Analyzer (M.E.A.D.)], Perfusion Index (PI) value of peripheral blood flow, and the changes of cortisol and IL-6 level in salivary fluid.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese or Taiwanese-proficient men and women aged ≥18 years.
2. Patients with stage I-III breast cancer.
3. Suffering from peripheral neuropathy caused by chemotherapy (professional judgment by a physician).
4. Willing to adhere to requirement that no new pain medication be taken throughout the study period.
5. Willing to adhere to all study-related procedures, including randomization to one of the two arms.
6. Patient answers "Yes" to at least one factor in the question: "Do participants think your balance, gait, posture, alignment, or flexibility has been affected by your experience of CIPN?"

Exclusion Criteria:

1. Metastatic disease.
2. Drugs abuse such as amphetamines, morphine, etc.
3. Pregnant
4. Those with severe mental illness or mental instability who cannot cooperate with the trial.
5. People who are severely hearing impaired, visually impaired, or demented and unable to perform yoga.
6. Severe heart disease or chronic obstructive lung disease, liver or kidney failure,and edema or severe skin damage.
7. Severe spinal disease, affecting actors.
8. Those who have participated in yoga practice in the past month.
9. Those who do not sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-12-21 (Actual)

PRIMARY OUTCOMES:
Neuropathic Pain Scale | Change from baseline of Neuropathic Pain Scale at 8 weeks.
  The questionnaire explores the performance of patients with neuropathic pain and nociceptive pain in different pain types in this questionnaire, and has appropriate reliability and validity, among which, specific pain performance, for different types of pain and changes in nerve conduction examination have special performance.
  This questionnaire is NPSI-T(Chinese version of neuropathic pain symptom inventory). It consists of 12 questions, all of which address pain on a scale of 0-10. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Peripheral perfusion index | Change from baseline Peripheral perfusion index at 8 weeks.
  The investigators expected to observe changes in peripheral perfusion values to reflect the correlation between peripheral blood flow and peripheral neuropathy.
  The normal value of Peripheral perfusion index(PPI) was suggested to range between 0.2 and 20%.Higher Peripheral perfusion index values reflects better peripheral tissue perfusion.

OTHER OUTCOMES:
Salivary Cortisol level | Change from baseline Salivary cortisol level at 8 weeks.
  Cortisol plays an important role in the energy metabolism, and is regarded as one of the main stress hormones.
Interleukin-6(IL-6) level | Change from baseline Salivary Interleukin-6(IL-6) level at 8 weeks.
  The investigators suggest that Interleukin-6(IL-6) signaling may be an important biological mechanism associated with the persistence of painful CIPN symptoms
Meridian Energy Analyzer | Change from baseline at 8 weeks.
  The investigators use the Meridian Monitoring System test to detect changes in the conductivity of the skin on the surface of the meridians, in order to judge the changes in the energy of the mWeeridians of the body.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University, Taiwan, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No